CLINICAL TRIAL: NCT03628547
Title: Assessment of Musculoskeletal Pain and Psychosocial Status of Professional and Amateur Athletes in Different Disciplines
Brief Title: Assessment of Musculoskeletal Pain and Psychosocial Status of Athletes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, amine atac, research assistant, Istanbul Medipol University Hospital
Other Study IDs: 10840098-604.01.01-E.30223
Record Dates: First submitted 2018-08-10; First posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Pain
Keywords: musculoskeletal system pain; athlete; psychosocial problems; algometer
MeSH Terms: conditions — Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- soccer players: Measuring devices and questionnaires will be applied to assess the pain and psychosocial states of musculoskeletal system of 10 amateur soccer players and10 professional soccer players.
  Interventions: Behavioral: Measuring devices and questionnaires
- basketball players: Measuring devices and questionnaires will be applied to assess the pain and psychosocial states of musculoskeletal system of 10 amateur basketball players and10 professional basketball players.
  Interventions: Behavioral: Measuring devices and questionnaires
- volleyball players: Measuring devices and questionnaires will be applied to assess the pain and psychosocial states of musculoskeletal system of 10 amateur volleyball players and10 professional volleyball players.
  Interventions: Behavioral: Measuring devices and questionnaires
- runners: Measuring devices and questionnaires will be applied to assess the pain and psychosocial states of musculoskeletal system of 10 amateur runners and 10 professional runners.
  Interventions: Behavioral: Measuring devices and questionnaires
- table tennis athlete: Measuring devices and questionnaires will be applied to assess the pain and psychosocial states of musculoskeletal system of 10 amateur table tennis athlete and 10 professional table tennis athlete.
  Interventions: Behavioral: Measuring devices and questionnaires
- field tennis athlete: 10 amateur field tennis athlete 10 professional field tennis athlete
  Interventions: Behavioral: Measuring devices and questionnaires
- kickboxers: Measuring devices and questionnaires will be applied to assess the pain and psychosocial states of musculoskeletal system of 10 amateur kickboxers and 10 professional kickboxers.
  Interventions: Behavioral: Measuring devices and questionnaires
- archers: Measuring devices and questionnaires will be applied to assess the pain and psychosocial states of musculoskeletal system of 10 amateur archers and 10 professional archers.
  Interventions: Behavioral: Measuring devices and questionnaires

INTERVENTIONS:
Behavioral: Measuring devices and questionnaires — Measuring devices and questionnaires will be applied to assess the pain and psychosocial states of musculoskeletal system of athletes. The Expanded Scandinavian Muscle Skeleton Questionnaire (NMQ) and Visible Analogue Scale (VAS) will be used to identify and assess the symptoms of musculoskeletal discomfort as 'pain'. The participant will be evaluated with the algometer, the sporty trust will be questioned with the Sporty Trust Continuous Inventory, and the Quality of Life will be assessed with the World Health Organization Quality of Life Scale Short Form and Depression will be evaluated with Beck Depression Inventory.

SUMMARY:
The sporty performance exhibited by an athlete faces physiological, biomechanical and psychological activity of the athlete. It depends on both the psychological state and the elevation of the musculoskeletal system to a certain level so that the athlete can perform optimally and excellently. For this reason, we aimed to evaluate the musculoskeletal system pain of amateur and professional athletes in different disciplines and the psychosocial states such as sports confidence, depression and quality of life.

DETAILED DESCRIPTION:
This study consists of 80 amateur and 80 professional sportsmen who are participating in sports by doing sports in soccer, basketball, volleyball, athletics, table tennis, field tennis, folk dances, kickboxing and archery branches between the ages of 15 and 36. The Expanded Scandinavian Muscle Skeleton Questionnaire (NMQ) and Visible Analogue Scale (VAS) will be used to identify and assess the symptoms of musculoskeletal discomfort as 'pain'. The participant will be evaluated with the algometer, the sporty trust will be questioned with the Sporty Trust Continuous Inventory, and the Quality of Life will be assessed with the World Health Organization Quality of Life Scale Short Form and Depression will be evaluated with Beck Depression Inventory.

ELIGIBILITY:
Inclusion Criteria:

* The athletes and their coaches must be voluntary and willing.
* During the evaluation, the athletes must give careful and relevant answers to the measuring instruments.
* They have to actively run the sport they belong to.

Exclusion Criteria:

* Having undergone a surgical operation due to sports injuries in the last 3 weeks
* The athletes do not want to answer the surveying instruments

Ages: 15 Years to 36 Years | Sex: All
Age Groups: Child, Adult
Study Population: Participants will be between the ages of 15 and 36
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2018-08-15 (Estimated); Primary Completion 2018-10-17 (Estimated); Study Completion 2018-12-03 (Estimated)

PRIMARY OUTCOMES:
Musculoskeletal system pain | 1 month
  Participants' musculoskeletal system pain will asses by using Nordic and algometer.

SECONDARY OUTCOMES:
Sporty confidence | 1 month
  Participants' sporty confidence will asses by using continuous sportive trust inventory.
Health Related Quality of Life | 1 month
  Participants' health Related Quality of Lifequality of life will asses by using World Health Organization Quality of Life Scale Short Form (WHOQOL-BREF)
Depression | 1 month
  Participants' depression will asses by using Beck Depression Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Şahin, Study Director — Medipol University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kahraman T, Genc A, Goz E. The Nordic Musculoskeletal Questionnaire: cross-cultural adaptation into Turkish assessing its psychometric properties. Disabil Rehabil. 2016 Oct;38(21):2153-60. doi: 10.3109/09638288.2015.1114034. Epub 2016 Jan 4. PMID 26726840
- [Result] Aghilinejad M, Choobineh AR, Sadeghi Z, Nouri MK, Bahrami Ahmadi A. Prevalence of Musculoskeletal Disorders among Iranian Steel Workers. Iran Red Crescent Med J. 2012 Apr;14(4):198-203. Epub 2012 Apr 1. PMID 22754681
- [Result] Wang YP, Gorenstein C. Psychometric properties of the Beck Depression Inventory-II: a comprehensive review. Braz J Psychiatry. 2013 Oct-Dec;35(4):416-31. doi: 10.1590/1516-4446-2012-1048. Epub 2013 Dec 23. PMID 24402217